CLINICAL TRIAL: NCT04439097
Title: Short and Medium-term Effects of a Multicomponent Physical Exercise Program With a Mediterranean Diet on Bone Mineral Density, Gait, Balance, and Fall Risk for Patients With Alzheimer's Disease: Randomized Controlled Clinical Trial Study Protocol
Brief Title: Effects of Multicomponent Physical Exercise Program and Mediterranean Diet in Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Roberto Méndez Sánchez, Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02102009-USalamanca
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Alzheimer Disease; Physical Exercise; Bone Density; Fall
MeSH Terms: conditions — Alzheimer Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is a randomized parallel-group, single blinded controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: will perform all evaluations without knowing the group to which the patients have been assigned, and they will not have a relationship with the physiotherapist who applies the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients allocated to the intervention group will perform a MPEP during 6 months, with a frequency of 3 sessions per week, and approximately 45-50 minutes of duration each session. In addition, they will have a Mediterranean Diet.
  The patients in the MPEP will be carried out in small groups of 5-8 people. Structure of sessions: 3 different parts: an initial warm-up, a main part and a final cool-down and relaxation.
  Interventions: Other: Multicomponent physical exercise program associated with a Mediterranean diet
- Control Group (Active Comparator): Participants allocated to the control group will receive usual care and continue with their life normally, without participating in a standardized exercise program. They will be instructed to maintain their current physical activity level.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Multicomponent physical exercise program associated with a Mediterranean diet — In this basic structure of each sessions, traditional exercises of mobility, strength, balance and coordination are included with the main objective of improving functional capacities. But, besides, games and some activities are also included with the aim, not only of improving the functional capacity, but also working the cognitive functions to reinforce the global effects.
  The Mediterranean diet will based in these main foods: 1) vegetables; 2) fruits; 3) fish or seafood; 4) legumes; 5) nuts; 6) bread or cereals; 7) white meat; 8) eggs; and 9)olive oil.
  Arms: Experimental Group
Other: Usual care — Usual care and participants continue with their life normally, without participating in a standardized exercise program, and they will be instructed to maintain their current physical activity level.
  Arms: Control Group

SUMMARY:
This study is a randomized, parallel-group, single blinded controlled clinical trial. The general objective of this multicomponent physical exercise program (MPEP) associated with a Mediterranean Diet (MeDi) is to decrease the risk of falls and fractures through the improvement of the bone health and physical functions of people with Alzheimer Disease.

Patients allocated to the intervention group will perform a MPEP with a MeDi during 6 months, with a frequency of 3 sessions per week, and approximately 45-50 minutes of duration each session.

During the study, 4 evaluations will be carried out to assess the effects of the interventions on bone mineral density, gait, balance, and fall risk: ((1) Baseline (pre-intervention); 2) 1st post-intervention after 1 month; 3) 2nd post-intervention after 3 months; 4) Final, 3rd post-intervention after 6 months

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes older than 50 years
* Have a diagnosis of AD
* Present mild or moderate cognitive impairment (Mini-mental State Examination (MMSE) score between 11 and 23 points included)
* Acceptance to participate in the study (enrollment in the study and signing of informed consent)

Exclusion Criteria:

* Other associated pathologies that do not allow physical exercise due to having severe functional disability or being insecure (neurological diseases, severe cardio-respiratory pathology, etc.).
* Impossibility to carry out the evaluation tests.
* Falls and other incidents with severe consequences that cause disability and/or that do not allow the intervention to continue.
* Attendance at the MPEP is less than 75% in the total of the sessions between assessments. (Criterion applied to each period between assessments).
* Not performing the MPEP sessions for 2 or more consecutive weeks.
* Participate in another intervention program outside of this study, especially an exercise program (important intervention bias for the control group).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in gait and balance 1 | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Tinetti's Performance Oriented Mobility Assessment (POMA-T) will be used (points). the original POMA-T 28-point version. It consists of a balance scale (Balance performance oriented mobility assessment (POMA-B) can score 16 points) and a gait scale (Gait performance oriented mobility assessment (POMA-G) can score 12 points )
Change in gait and balance 2 | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Timed up and go test (TUG) will be used (s). IT measures the time in seconds for the subjects to get up from a standard armchair, walk 3 metres, turn, walk back to the chair and sit down. The cut-off point for normal mobility is 12 seconds and values > 30 s indicate a high level of dependence. (a time <10s it is considered normal; <20s mobility difficulties and low or moderate risk of falls; > 20 mobility problems with need of help and high risk of falls)
Change in Bone Mineral Density (BMD) | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Bone health status will be assessed by ultrasound calcaneus densitometry/sonometry. As primary outcome we will assess the estimated BMD (g/cm2).
Change in T-Score as primary parameter of bone health | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Bone health status will be assessed by ultrasound calcaneus densitometry/sonometry. As primary outcome we will assess the T-Score. A T-score shows how much the BMD is higher or lower than the BMD of a healthy 30-year old adult. (-1.0 or above normal BMD; From -1.0 to -2.5 low BMD or osteopenia; -2.5 or below very low BMD and diagnosis of osteoporosis.

SECONDARY OUTCOMES:
Change in static balance | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  one-leg balance test (OLB) will be used (s). This test assess the ability of the patients to remain upright on one leg without support for at least 5 seconds, and each leg was tested.
Change in proactive balance | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Functional reach test (FR) will be used (cm). Is a measure of the distance in centimeters that the standing participant is able to reach forward from an initial upright posture to the maximal anterior leaning posture without moving or lifting the feet.
Falls during the study | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  The number of falls of each subject during the study will be counted
Change in the Broadband ultrasound attenuation (BUA) as secondary parameter of bone health | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Bone health status will be assessed by ultrasound calcaneus densitometry/sonometry. As secondary outcome we will assess the Broadband ultrasound attenuation (BUA) (dB/MHz). It is a measurement of the differential attenuation of sound waves transmitted through the calcaneus.
Change in the Speed of sound (SOS) as secondary parameter of bone health | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Bone health status will be assessed by ultrasound calcaneus densitometry/sonometry. As secondary outcomes we will assess the SOS through the calcaneus bone (m/s). It is calculated as the ratio of the distance traveled by the impulse and the time taken by the signal to travel that distance
Change in the Quantitative ultrasound index (QUI) as secondary parameter of bone health | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Bone health status will be assessed by ultrasound calcaneus densitometry/sonometry. As secondary outcomes we will assess the Quantitative ultrasound index. To improve precision we will calculate de QUI, a variable derived from the mathematical combination of both SoS and BUA [0.41 × (BUA + SoS) - 571] (19), expressed as percent.
Change in the nutritional status | 6 months. 4 time points: 1) Baseline (pre-intervention); 2) 1st post-intervention (1 month); 3) 2nd post-intervention (3 months); 4) Final, 3rd post-intervention (6 months)]
  Nutritional status will be assessed by the Mini Nutritional Assessment (MNA) (points). Total score ranging from 0 to 30. Well nourished (MNA score >23.5), at risk of malnutrition (MNA score=17.0-23.5), or malnourished (MNA score <17).

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Méndez-Sánchez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puente-Gonzalez AS, Sanchez-Gonzalez F, Hernandez-Xumet JE, Sanchez-Sanchez MC, Barbero-Iglesias FJ, Mendez-Sanchez R. Short and medium-term effects of a multicomponent physical exercise program with a Mediterranean diet on bone mineral density, gait, balance, and fall risk for patients with Alzheimer disease: Randomized controlled clinical trial study protocol. Medicine (Baltimore). 2020 Sep 18;99(38):e22385. doi: 10.1097/MD.0000000000022385. PMID 32957420